CLINICAL TRIAL: NCT01934413
Title: Technology-enhanced Transitional Care for Rural Palliative Care Patients: A Pilot Study
Acronym: TPC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Diane Holland, Clinical Nurse Researcher, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 13-006242
Record Dates: First submitted 2013-08-29; First posted 2013-09-04 (Estimated); Last update posted 2015-02-16 (Estimated); Status verified 2015-02

CONDITIONS: Palliative Care; Transitional Care
Keywords: Palliative Care; Technology; Rural; Transitional Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Technology-Enhanced TPC (Active Comparator): In addition to receiving usual palliative care service in the hospital setting, Technology-Enhanced Transitional Palliative Care patients will receive Transitional Care from the Palliative Care consulting team beginning in the hospital within 24 hours of study enrollment and continuing post discharge for eight weeks in their homes in rural locations by means of video visits with the Palliative Care consulting team.
  Interventions: Behavioral: Technology-Enhanced Transitional Palliative Care
- Usual standard of care (Other): The control group will receive only the current standard palliative care service in the hospital setting, which includes standard in-hospital palliative care consultation and standard discharge planning.
  Interventions: Other: Usual Standard of Care

INTERVENTIONS:
Behavioral: Technology-Enhanced Transitional Palliative Care — The Transitional Care intervention will be initiated within 24 hours after enrollment, and will include initial transitional care planning, daily hospital visits, crisis prevention planning by an experienced Palliative Care nurse. The intervention will continue after the patient is discharged to home or short term skilled nursing facility, and it will involve an in-person visit between 24-48 hours post discharge, weekly virtual visits via iPad and video conference technology, and additional home visits as needed. Care plans established during initial planning will be implemented and adjusted under the guidance of the palliative care nurse delivering the intervention.
  Arms: Technology-Enhanced TPC
Other: Usual Standard of Care — Usual care includes routine hospital discharge planning and usual physician care in primary and specialty outpatient clinics post hospital discharge. The PC consulting service provides consulting services in the inpatient setting. There are no standardized, intentional services provided to outpatients by the PC consulting team. Services provided to outpatients may occur sporadically as initiated by the patient. The majority of PC follow-up if any is a single phone call to the patient/caregiver. To account for the time spent and number of contacts made with the intervention group, the control group will be contacted by phone weekly by a non-nurse member of the study team not involved with the intervention, asked to relate what, if any, medically-related events occurred.
  Arms: Usual standard of care

SUMMARY:
The purpose of this pilot study is to develop and test a technology-enhanced transitional palliative care (TPC) intervention for patients and caregivers living in rural locations. The investigators hypothesize that access to palliative care will be improved, thereby improving patient and caregiver reported outcomes and decreasing the use of costly health services.

DETAILED DESCRIPTION:
The purpose of the proposed research is to design and evaluate a technology enhanced transitional palliative care (TPC) intervention for patients living in rural locations. The contributions of the proposed research are expected to address the gap in palliative care services and transitions of care for rural patients. This research is significant because it addresses the challenges of three independently important health care foci - needs of rural patients, care transitions, and the evolving field of palliative care. The study will not simply address the critical barrier imposed by distance, but also extend PC practice by improving transition management for the impending dramatic increase in seriously ill and dying patients in rural areas through evolving demographic shifts. The goal of the proposed research is to advance the development of transitional care strategies for rural PC patients and caregivers, and provide evidence of new ways to support continuity of care for patients with life-limiting conditions.

The study is guided by the "Transitional Care Model" or "TCM" as developed by Naylor which combines quality, cost, and satisfaction. The TCM has a solid evidence base from more than 15 years of multidisciplinary research. Unique features of the model include care that is delivered and coordinated by the same nurse across hospital and home settings 7 days per week for an average of 2 to 3 months using evidence-based protocols with a focus on long term outcomes. Core components of the model include a holistic, person/family centered approach and protocol guided care. The nurse functions as part of an interdisciplinary team with shared accountability, however, the nurse is the single "point person" across an episode of care providing the vital link from hospital to home. Inherent within the model is shared communication systems that span care settings.

A randomized control trial design will be used. Community dwelling adult patients and their caregivers who receive a palliative care consult while hospitalized in the hospital will be enrolled in the study, then randomized to group membership and followed for a total of 8 weeks after hospital discharge. Following a detailed protocol for TPC, the intervention group will receive weekly video session visits (using computer software that allows audio/visual contact through the computer screen) by the study nurse. The investigators will determine the feasibility and acceptability of the TPC intervention and study methods and procedures when engaging palliative care patients and their caregivers. The investigators will compare patient and caregiver reported outcomes and determine effect size for patients receiving technology-enhanced TPC (intervention group) to patients in the control group, and they will explore the impact of the technology-enhanced TPC intervention on health care service utilization.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients hospitalized at study site, and their designated caregiver (if available)
* Receiving palliative care
* Returning home or to a facility for short term (30 days) rehabilitation
* Able to provide informed consent
* Able to complete self-reported questionnaires without assistance

Exclusion Criteria:

* Long-term placement in skilled nursing facility after hospitalization
* Receiving hospice
* Living within city limits of hospital
* Cognitive impairments
* Non-English speaking

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2013-09; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Change in mean scores on FACIT-Pal Questionnaire | Baseline, 1 month post-enrollment, 2 months post-enrollment
  The patient's quality of life will be determined by the change in mean scores from baseline to 1 month and 2 months post enrollment, using the Functional Assessment of Chronic Illness Therapy - Palliative Care Scale (FACIT-Pal). The FACIT-Pal palliative subscale contains 19 questions specific to persons with life-limiting illness. Each item is rated on a 5 point numeric rating scale from 9 (not at all) to 4 (very much). Scores range from 0-76. Higher scores indicate better quality of life.

SECONDARY OUTCOMES:
Change in mean scores on ESAS-r Questionnaire | Baseline, 1 month post-enrollment, 2 months post-enrollment
  The patient's symptom intensity will be determined by the change in mean scores from baseline to 1 month and 2 months post enrollment, as measured by the Edmonton Symptom Assessment System (revised) ESAS-r scale, The ESAS-r captures the patient's perspective on 9 symptoms that are common in palliative care (pain, tiredness, drowsiness, nausea, lack of appetite, shortness of breath, depression, anxiety, wellbeing). An optional 10th symptom can be reported. Each symptom is rated on an 11 point numeric rating scale from 0 (symptom absent or best) to 10 (worst possible). Scores range from 0-100, with lower scores indicating patient perceives fewer or no symptoms and higher scores indicating patient perceives worse symptoms.

OTHER OUTCOMES:
Health Care Service Utilization | Baseline to 6 months after enrollment
  Health Services information will be summarized by review of medical records and administrative databases for number of unplanned hospitalizations, number of intensive care unit days, total length of hospital stay (days), number of emergency department visits, number of clinic office visits, number of home healthcare visits, time (in days) to hospice admission, and time (days) receiving hospice.

CONTACTS AND LOCATIONS:
Overall Officials: Diane E Holland, PhD, RN, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Health System, Mankato, Minnesota, United States